CLINICAL TRIAL: NCT04925115
Title: Effect of Physical Activity on Academic Stress While Controlling the Confounding Variables
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/00930 Salman khan
Record Dates: First submitted 2021-03-12; First posted 2021-06-14 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Stress

STUDY DESIGN:
Intervention Model Description: Two groups with randomization, Assignment: Brisk walking
Who Masked: Participant
Masking Description: According to study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Interventional group:
  1. Warm up and cool down (10 minutes before physical activity)
  2. Brisk walking ( 30 minutes each session for 5 days in a week)
  3. Week 1 to week 6 same protocol
  Interventions: Other: Brisk walking
- Control group (No Intervention): Routine activity of daily life

INTERVENTIONS:
Other: Brisk walking — * Warm up and cool down (10 minutes before physical activity)
  * Brisk walking ( 30 minutes each session for 5 days in a week)
  Other Names: Moderate physical activity
  Arms: Interventional group

SUMMARY:
The study is designed to determine the effectiveness of moderate physical activity on academic stress with controlling and observing on confounding variables.

DETAILED DESCRIPTION:
Now a days, modern time, new researches increased knowledge of researchers on physical activity and its effect on academic stress. Literature search shows to reduce academic stress among people all types of physical activities were effective and useful. Particularly moderate level of physical activity like brisk walking was significantly associated with academic stress, as compare to hard and light physical activities. Many Studies and research was available on the effectiveness of physical activities and found effective for dealing with academic stress but these were single centered and lacking control on confound variables observation, For example, Age, BMI, Socio-economic status, Semester pressure, Curriculum burden, depression, anxiety ,stress , demographics etc were absent in previous studies plus the available research is partial, includes only females. This research will be impartial and free from gender discrimination. Both male and female students will be taken in consideration for test and a multi-centered study will be conducted focusing on the confounding variables to determine the effectiveness of physical activity on academic stress with controlling variables is the recommendation of this research

ELIGIBILITY:
Inclusion Criteria:

* Participants falling in this category would be recruited into the study.
* Moderate academic stress

Exclusion Criteria:

* Participant falling in this category would be excluded from the study.
* Physical Disability
* Acute infection
* Chronic infection
* Acute inflammation
* Chronic inflammation
* Known osteoporosis
* Individual with respiratory diseases e.g. asthma
* Smoking
* Musculoskeletal injuries

Confounding variables:

* Age
* Gender
* BMI
* Socio-economic status
* Semester
* Depression, anxiety and stress
* Demographic (rural, urban)
* Relationship status (married and unmarried)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Estimated)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Academic Stress scale | 6 weeks
  Academic Stress will be measured through 40 item scale (Academic Stress scale). It will be used during survey for inclusion criteria, This scale consists of 40 items describing the stress in your institution/ college life from the various sources.
Perceived stress scale | 6 weeks
  Perceived stress scale will be measured through 10 questions in this scale ask you about your feelings and thoughts during the last month. In each case, you will be asked to indicate by circling how often you felt or thought a certain way. As 0 = Never 1 = Almost Never 2 = Sometimes 3 = Fairly Often 4 = Very Often
Depression, Anxiety and Stress Scale (DASS21) | 6 weeks
  Depression, anxiety and stress scale will be measured through 21 items scale. Moderate stress score is : 19-25
Physical Activity Readiness Questionnaire (PAR-Q) | 6 weeks
  Physical Activity Readiness Questionnaire (PAR-Q)
  Yes to one or more questions:
  If you have not recently done so, consult with your doctor by telephone or in person before increasing your physical activity and/or taking a fitness appraisal. Tell your doctor what questions you answered 'yes' to on PAR-Q or present your
  PAR-Q copy. After medical evaluation, seek advice from your doctor as to your suitability for:
  Unrestricted physical activity starting off easily and progressing gradually, and Restricted or supervised activity to meet your specific needs, at least on an initial basis.
  If you answered PAR-Q accurately, you have reasonable assurance of your present suitability for:
  A graduated exercise programme A fitness appraisal

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No